CLINICAL TRIAL: NCT00306956
Title: Influence of Pacifiers on Breastfeeding Duration: a Multicentre, Randomised Controlled Trial
Brief Title: Influence of Pacifiers on Breastfeeding Duration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Salud Materno Infantil (Other)
Collaborators: International Childrens Medical Research Association, Switzerland. (Unknown)
Responsible Party: Alejandro Jenik, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: FUNDASAMIN101
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Sudden Infant Death
Keywords: Infant; Newborn; pacifier; dummies; breastfeeding; Sudden Infant Death; SIDS; Pacifiers
MeSH Terms: conditions — Sudden Infant Death; Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Recommendation to offer a pacifier to 15 days old newborn infants with successful breastfeeding
  Interventions: Behavioral: offer a pacifier
- B (Active Comparator): Recommendation not to offer a pacifier to normal newborn infant with successful breastfeeding at 15 days of age
  Interventions: Behavioral: offer a pacifier

INTERVENTIONS:
Behavioral: offer a pacifier — To offer a pacifier to normal newborn infants at 15 days of age

SUMMARY:
The purpose of this study is to determine if the introduction of pacifier use to infants at 2 weeks of age, once breast feedings are well established, will affect the incidence and duration of successful breastfeedings.

DETAILED DESCRIPTION:
The incidence of Sudden infant death syndrome in developing countries is comparable with that of developed countries. Two important risk factors with implications for prevention are prone sleeping position and the association with smoke. Also, breastfeeding has been reported to be protective against SIDS.

In accordance with WHO/UNICEF recommendations, lactation consultants and other health professionals within "Baby-Friendly" institutions typically discourage the use of pacifiers in breastfed infants. The recent American Academy of Pediatrics policy statement, however, recommends pacifier use, during periods of sleep as a potential method to reduce the risk of SIDS. Previous observational studies had been unanimous in reporting an approximate doubling of the risk of early weaning with daily pacifier use. However, randomized controlled trials in developed countries, have not shown that giving pacifiers results in shorter breastfeeding duration, except when pacifiers are given in the first 5 days. It has therefore been seen that practically every author of a major study on the association between breastfeeding and pacifier use has proposed that the question can only be fully and completely answered by randomized studies. To date there are no large randomized studies evaluating the influence of pacifier use on breastfeeding duration.

Our Primary outcome is to compare the prevalence of exclusive breastfeeding at three months in infants between groups randomised to pacifier and no pacifier exposure once breastfeedings have been fully established.

Second outcome: to evaluate the effects of the pacifier's introduction when breastfeeding is firmly established at 15 days on the duration of breastfeeding.

Recruitment to the trial will take place in several public and private hospitals.

Those mothers who do not show a strong preference in regards to the introduction of the pacifier, will be randomised during the postpartum visit at 2 weeks (if well established breastfeeding is present) on two arms:

1. No pacifier,
2. Pacifier introduced at 15 days.

Structured telephone interviews will be conducted at 1, 2, 3, 4, 5, and 6 months and every 60 days thereafter until the breastfeeding has ended to record breastfeeding duration and type (exclusive or not) and pacifier use.

ELIGIBILITY:
Inclusion Criteria:

The following patients will be invited to participate before hospital discharge:

* Women who agree not to introduce the pacifier before 2 weeks
* Intention to exclusively breastfeed their infants for at least 3 months
* Breastfeeding exclusively at discharge
* Delivered a healthy singleton newborn
* 37 completed weeks and at least a 2.5 kg birth weight
* Possibility of contact by telephone
* Patients will be randomized at age 15 days if:

  * They are exclusively breastfeeding
  * They have no existing breastfeeding problems
  * Babies use no pacifiers.
  * Breastfeeding is well established
  * No maternal risk factors for lactation problems

Exclusion Criteria:

* Extremely or persistently sore nipples
* Presence of mastitis or abscess formation.
* Medical situations contraindicating breastfeeding

Ages: 14 Days to 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1021 (Actual)
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The prevalence of exclusive breastfeeding for three month old infants between groups randomised to pacifier and no pacifier exposure. Pacifier introduction is delayed until 15 days to ensure that breastfeeding is firmly established. | Three months

SECONDARY OUTCOMES:
To evaluate the effects of the pacifier's introduction when breastfeeding is firmly established at 15 days on the duration of breastfeeding | one year
To evaluate the median breastfeeding duration in months in relation to the frequency of pacifier use | one year
To test whether pacifier use is causally related with muguet, otitis and sore nipples | one year
Compliance with group assignment | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Jenik, M.D., Principal Investigator — Jefe de Recién Nacido Normal, Hospital Italiano, Buenos Aires
Locations (5):
- Argentina (5):
  - Hospital Privado del Sur, Bahía Blanca, Buenos Aires
  - Hospital Diego Paroissien, Isidro Casanova, Buenos Aires
  - Hospital Municipal Materno Infantil de San Isidro "Dr. Carlos Gianantonio", San Isidro, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Sanatorio de la Trinidad, Buenos Aires